CLINICAL TRIAL: NCT02762357
Title: Post-Marketing Clinical Follow-up (PMCF) Study to Evaluate the Safety and Efficacy of Novosyn® Quick Suture Material for Episiotomy . A Monocenter, Prospective, Observational Study.
Brief Title: PMCF-study Using Novosyn® Quick Suture Material for Perineal Repair After Episiotomy
Acronym: EPINOQ
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1504
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Episiotomy
Keywords: Novosyn Quick; Episiotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Novosyn® Quick: episiotomy closure using suture material
  Interventions: Device: Novosyn® Quick

INTERVENTIONS:
Device: Novosyn® Quick — Episiotomy closure

SUMMARY:
The aim of this study is to show that the performance of Novosyn® Quick suture material is comparable with other suture material used for episiotomy. In order to show that, various safety and efficacy parameters have been selected. The outcome regarding these parameters will be evaluated by a quantitative summary of the available clinical data from the literature. Study population consists of women with a spontaneous vaginal delivery who required perineal repair due to an episiotomy.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women who require perineal repair due to an episiotomy after spontaneous vaginal delivery.
* Singleton birth between 37 and 42 weeks gestation
* Written informed consent

Exclusion Criteria:

* Age< 18 years
* Previous perineal surgery
* Instrumental vaginal deliveries
* Multiparous (at least 1 previous perineal delivery)
* Episiotomy involving the anal sphincter or the rectum
* Medical consumption that might adversely affect healing
* Women with active infection at the time of delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Incidence of wound dehiscence | 3 months postpartum
  A dehiscence of the skin which needs surgical treatment with re-closure.

SECONDARY OUTCOMES:
Incidence of Re-suturing | 3 months postpartum
  Re-suturing due to wound dehiscence
Incidence of suture removal | 3 months postpartum
  Suture removal due to wound problems (infection, gaping wound, residual material requiring removal)
Short-term perineal pain (VAS) | 24h to 48h, 10 days postpartum
Long term perineal pain (VAS) | 3 months postpartum
Pain in daily living (VAS) | 24h and 10 days postpartum
  Pain in repose, during walking, during sitting, when urinating, and when defecating
Dyspareunia | 3 months post-operatively
  Questionnaire
Sexual intercourse | 3 months post-operatively
  Questionnaire
Patient satisfaction with the repair (VAS) | until 3 months postpartum

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General de Granollers, Granollers
  - IDC Hospital General de Catalunya, Sant Cugat Del Vallés

IPD SHARING:
Plan to Share IPD: No